CLINICAL TRIAL: NCT02398734
Title: Risk Reduction of Symptomatic and Silent Brain Infarctions During Carotid Endarterectomy by the Ultrasound Activation of Endogenous Fibrinolytic System Using Sonolysis (Transcranial Doppler Monitoring)
Brief Title: SONOlysis in Prevention of Brain InfaRctions During Internal Carotid Endarterectomy
Acronym: SONOBIRDIE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Ostrava (Other)
Collaborators: Ústřední fakultní vojenská nemocnice, Praha, Czechia (Unknown); Vítkovická nemocnice, Ostrava, Czechia (Unknown); Masarykova nemocnice v Ústí nad Labem, Ústí nad Labem, Czechia (Unknown); Nemocnice České Budějovice, České Budějovice, Czechia (Unknown); Fakultní nemocnice Hradec Králové, Hradec Králové, Czechia (Unknown); Fakultní nemocnice Plzeň, Plzeň, Czechia (Unknown); Krajská nemocnice Liberec, Liberec, Czechia (Unknown); Fakultná nemocnica Martin, Martin, Slovakia (Unknown); Nemocnice Jihlava, Jihlava, Czechia (Unknown); Nemocnice na Homolce, Praha, Czechia (Unknown); Fakultní nemocnice Motol, Praha, Czechia (Unknown); Fakultná nemocnica Nitra, Nitra, Slovakia (Unknown); Fakultní nemocnice Olomouc, Olomouc, Czechia (Unknown); Fakultná nemocnica Košice, Košice, Slovakia (Unknown); Krajská nemocnice T. Bati, Zlín, Czechia (Unknown); Allgemeine Krankenhausl Linz, Linz, Austria (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CZ20150305
Record Dates: First submitted 2015-03-20; First posted 2015-03-25 (Estimated); Last update posted 2022-12-06 (Actual); Status verified 2022-12

CONDITIONS: Internal Carotid Artery Stenosis
Keywords: sonolysis; carotid endarterectomy; stroke prevention; brain infarction
MeSH Terms: conditions — Carotid Stenosis; Brain Infarction

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sonolysis (Experimental): In patients randomized into sonolysis group, middle cerebral artery segment in a depth of 55 mm will be continuously monitored during intervention using a diagnostic 2-MHz transcranial Doppler probe with a maximal diagnostic energy. The probe will be fixed in a required position using a special helmet and sonolysis will start before the carotid intervention and will be stopped after the intervention, but at latest after 120 minutes. Transcranial Doppler machine with a 2-MHz diagnostic transcranial Doppler probe will be used. This non-diagnostic transcranial Doppler monitoring will be performed without detection of microembolic signals or detection of changes in blood flow. Device sound and Doppler wave imaging will be switched off. Only sonographer will be unblinded to the procedure.
  Interventions: Device: sonolysis
- Shame sonolysis (Sham Comparator): In patients randomized into control group, the transcranial Doppler probe will be fixed in a required position using a special helmet as in sonolysis group patients, but middle cerebral artery segment in a depth of 55 mm will be only localized using a diagnostic 2-MHz transcranial Doppler probe with a maximal diagnostic energy and the transcranial Doppler monitoring will be stopped afterwards. Patients in the control group will undergo a sham procedure in which further sonolysis (transcranial Doppler monitoring) will not be conducted.
  Interventions: Device: sonolysis

INTERVENTIONS:
Device: sonolysis — Continual transcranial Doppler monitoring of ipsilateral middle cerebral artery using a transcranial Doppler systems (e.g. DWL Multi-Dop T1, DWL, Sipplingen, Germany) with a diagnostic 2-MHz probe.
  Other Names: sonothrombolysis

SUMMARY:
SONOBIRDIE Trial is a randomized, single-blind, sham-controlled study designed for a demonstration of the safety and effectiveness of sonolysis (continual transcranial Doppler (TCD) monitoring) in reduction of risk of stroke or transient ischemic attack (TIA), brain infarctions and cognitive decline using a 2-MHz diagnostic probe with a maximal diagnostic energy on the reduction of risk of brain infarctions by the activation of endogenous fibrinolytic system during carotid endarterectomy (CEA) in patients with ≥ 70% symptomatic or asymptomatic internal carotid artery stenosis.

The sample size is based on an expected 2.5% reduction of ischemic stroke, TIA, and death during the 30-day postoperative period in the sonolysis group (estimated prevalence, 1.5 %) compared to the control group (estimated prevalence, 4 %). Pre-study calculations showed that a minimum of 746 patients in each group is needed to reach a significant difference with an alpha value of 0.05 (two-tailed) and a beta value of 0.8 assuming that 10 % would be lost to follow-up or refuse to participate in the study.

Consecutive patients will be assigned to the sonolysis or control group by a computer-generated 1:1 randomization. In patients randomized into sonolysis group, middle cerebral artery segment in a depth of 55 mm will be continuously monitored during intervention using a diagnostic 2-MHz TCD probe with a maximal diagnostic energy.

In patients randomized into control group, the TCD probe will be fixed in a required position using a special helmet as in sonolysis group patients, but middle cerebral artery segment in a depth of 55 mm will be only localized using a diagnostic 2-MHz TCD probe with a maximal diagnostic energy and the TCD monitoring will be stopped afterwards.

Confirmation of the investigators hypothesis that sonothrombolysis is able to activate endogenous fibrinolytic system during CEA with consecutive reduction of ischemic stroke, TIA or death, and the number and volume of brain infarcts, can lead to the increase of the safety of CEA in patients with internal carotid artery stenosis. The investigators can presume that up to 50% of patients indicated for CEA can be treated using these methods in the future.

DETAILED DESCRIPTION:
Results of the NASCET, ECST and ACAS studies showed that carotid endarterectomy (CEA) was a beneficial therapy for patients with a symptomatic internal carotid artery (ICA) stenosis >50% and asymptomatic ICA stenosis >60%, resp. Surgical risk of CEA varied between 2 and 15 % and even clinically silent microembolism can cause microinfarctions presenting with postoperative cognitive deficit.

Transcranial Doppler (TCD) monitoring during CEA is a common diagnostic method being used for the detection of microemboli and changes of blood flow in intracranial arteries. Reduction of periprocedural complications of CEA with TCD monitoring referred in some studies should be not only due to sophisticated indication of shunt implementation, optimization of surgery and anesthesia but also due to TCD activation of endogenous fibrinolytic system (equal to sonothrombolysis in acute stroke studies). Recently published SONOBUSTER Trial showed that intraoperative sonolysis reduced both the incidence and the volume of new brain infarctions following CEA.

There are 2 possible effects of ultrasound on thrombus - mechanical destruction due to vibration of thrombus with acceleration of penetration of fibrinolytics into thrombus and elevation of temperature and stimulation of endothelium with local activation of fibrinolytic system. Grant project NR/9487-3/2007 showed that TCD monitoring has a significant effect on activation of fibrinolytic system in healthy volunteers.

STUDY OBJECTIVES The objective of the randomized, double-blind, sham-controlled study is to demonstrate the safety and effectiveness of sonolysis (continual TCD monitoring) using a 2-MHz diagnostic probe with a maximal diagnostic energy on the reduction of stroke, transient ischemic attack (TIA) and brain infarction by the activation of endogenous fibrinolytic system during CEA in patients with ≥70% symptomatic or asymptomatic ICA stenosis.

The substudy aims to compare the risk of brain infarction detected using magnetic resonance between sonolysis and control group.

STUDY DESIGN

Overview:

SONOBIRDIE Trial is a randomized, single-blind, sham-controlled study designed for a demonstration of the safety and effectiveness of sonolysis (continual TCD monitoring) in reduction of risk of ischemic stroke, TIA, death, brain infarctions and cognitive decline by the sonolysis during CEA in patients with ≥70% ICA stenosis.

Expected sample size:

The sample size is based on an expected 2.5% absolute risk reduction of ischemic stroke, TIA and death during the 30-day postoperative period in the sonolysis group (estimated prevalence, 1.5%) compared to the control group (estimated prevalence, 4%). Pre-study calculations showed that a minimum of 746 patients in each group is needed to reach a significant difference with an alpha value of 0.05 (two-tailed) and a beta value of 0.8 assuming that 10% would be lost to follow-up or refuse to participate in the study.

The sample size for substudy is based on an expected 15% reduction of new ischemic lesions on diffusion weighted imaging-MRI (DWI-MRI) in the sonolysis group (estimated prevalence, 10%) compared to the control group (estimated prevalence, 25%). Pre-study calculations showed that a minimum of 112 patients in each group was needed to reach a significant difference with an alpha value of 0.05 (two-tailed) and a beta value of 0.8 assuming that 10 % would be lost to follow-up or refuse to participate in the study.

Test device:

The transcranial Doppler systems (e.g. DWL Multi-Dop T1, DWL, Sipplingen, Germany) with a diagnostic 2-MHz probe will be used for sonolysis (non-diagnostic TCD Doppler monitoring).

Sonolysis:

In patients randomized into sonolysis group, MCA segment in a depth of 55 mm will be continuously monitored during intervention using a diagnostic 2-MHz TCD probe with a maximal diagnostic energy (TIC~1.3), sample volume 10 mm.

Sham procedure:

In patients randomized into control group, the TCD probe will be fixed in a required position using a special helmet as in sonolysis group patients, but MCA segment in a depth of 55 mm will be only localized using a diagnostic 2-MHz TCD probe with a maximal diagnostic energy and the TCD monitoring will be stopped afterwards.

Carotid endarterectomy:

Surgery will be performed in a general or a local anesthesia (decision will be left to the discretion of the operating team) using a cut in front angle of the sternomastoid muscle. Common carotid artery (CCA) and later ICA and external carotid artery (ECA) will be cut free. Common carotid artery, ICA and ECA will be temporarily closed. Using a longitudinal cut of CCA and ICA, atherosclerotic plaque will be visualized. Plaque will be withdrawn under the microscopic control and later a suture of arteriotomy will be performed using a monophil non-absorbent fibre 6/0. Just before the end of surgery, haemostatic process will be controlled and drainage will be done. Surgery will be completed by suture of subcutis and cutis. Unfractioned heparin (100 IU/kg bodyweight) will be administered in all patients just before the arteriotomy. In the case of the insufficient collateral flow into MCA after clipping of the CCA and ICA, a temporal shunt will be used. Antiplatelet therapy (Aggrenox, clopidogrel 75 mg/day or acetylsalicylic acid 100 mg/day) will be used continuously in all patients. Surgeon will be blinded to sonolysis or sham procedure.

Magnetic resonance imaging:

Magnetic resonance imaging will be performed in patients enrolled to the substudy. Magnetic resonance imaging protocol consists of 4 sequences: 1. T2TSE; 2. DWI. Sequences 1 - 3 will be applied in the same level, they will have the same slice thickness and the same cut number. The slice thickness comprises its own cut thickness (5 mm) + distant factor (30 %). Standard number of slices will be 19. Standard slice level is considered to be a modified level of skull base due to the minimalization of distant artifacts. Diffusion weighted sequence shows a middle (average) diffusivity of every point of the examined brain tissue when b value is 500 and 1000. This sequence is applied in order to assess hemorrhage (T2*EPI) and to monitor sites of the reduced diffusion (DWI, b=500 and 1000); 3. T2 star-weighted gradient-recalled echo (GRE) sequence for detection of bleeding (including microbleeds); 4. Fluid-attenuated inversion recovery (FLAIR). Presence of new infarctions will be evaluated separately in the whole brain, in the intervened ICA territory and in the contralateral ICA territory.

New ischemic lesions in the brain are defined as hyperintense lesions on postintervention DWI sequences which were not present on the pretreatment MRI.

The volume of new brain infarctions will be measured manually. Ischemic lesions in the brain will be evaluated by two blinded investigators by consensus.

Clinical examinations and cognitive tests:

Standard physical and neurologic examinations (including the National Institutes of Health Stroke Scale - NIHSS, modified Rankin scale - mRS, and Addenbrooke's Cognitive Examination Revised - ACE-R) will be performed prior to CEA, 24 hours after CEA, 30 days and 1 year after randomization.

Randomization:

Consecutive patients will be assigned to the sonolysis or control group by a computer-generated 1:1 randomization.

ANALYSIS SETS

Efficacy analyses will be performed primary for the intent-to-treat population. The secondary analysis will be performed also for per-protocol population. The intent-to-treat population will consist of all randomized subjects who signed informed consent. The per-protocol population will exclude all subjects in the intent-to-treat population who did not have any major protocol deviations:

* Violation of inclusion or exclusion criteria.
* Withdrawal of consent within 30 days
* Crossing-over to the other treatment arm. Cross-overs are defined as patients randomized to the control group who receive continuous TCD monitoring for 10 minutes or longer and patients randomized to the sonolysis group who receive less than 10 min of sonolysis.
* Total time of sonolysis less than 40 min for patients randomized to the sonolysis group
* Total time of TCD monitoring of 40 min or more for patients randomized to the control group
* Carotid endarterectomy not within 2 days (48 hours) of randomization
* Not attending at least one of visits 3 (24 hours after CEA), 4 (30 days after CEA), or 5 (1 year after CEA)
* Outcomes assessed outside the specified time windows

The safety population consists of all subjects in the FAS who did receive one of the study interventions. Subjects will be analyzed according to the treatment they actually received (as treated):

* Patients randomized to the control group who receive continuous TCD monitoring for 10 minutes or longer will be considered to have received sonolysis.
* Patients randomized to the sonolysis group who receive less than 10 min of sonolysis will be considered to have received the control intervention.

STATISTICAL METHODS The primary analysis will be based on the full analysis set. Missing data will be handled according to Statistical Analysis Plan. The proportion of the composite of ischemic stroke, TIA, or death within 30 days will be calculated in both groups with a 95% Wilson score confidence interval. Groups will be compared using the chi-squared test. As an effect measure we will calculated the absolute risk difference with Newcombe hybrid score 95% CIs.

Mortality will be graphically depicted by Kaplan-Meier curves for each treatment group. Groups will be compared using a log-rank test. Mortality at 30 days for both groups and the difference between groups will be calculated with 95% CI from the Kaplan-Meier estimator. A risk difference with 95% CI will be provided, calculated on the log-scale using Greenwood standard errors and a normal approximation.

The proportion of any stroke and myocardial infarction within 30 days will be calculated for each group using the non-parametric cumulative incidence function estimator with death as competing event and 95% CI. Changes in cognitive functions will be compared between groups using a linear regression with baseline values and the group as covariates (usually referred to as ANCOVA). Assumptions for linear regression (homoscedasticity and normality of the errors) will be verified using residual-vs-fitted and QQ-plots. If the assumptions are not met, transformations (e.g. log), more robust methods (e.g. robust standard errors) or non-parametric methods will be considered.

Binary substudy outcomes (appearance of at least one new lesion) will be compared using chi-squared tests. The effects will be presented as absolute risk differences with Newcombe hybrid score 95% CIs.

The number of new lesions will be compared between groups using an exact Poisson test. The effect will be presented as incidence rate ratio with an exact 95% CI.

Multivariable logistic regression analyses will be used to analyze possible predictors of the primary outcome (composite of ischemic stroke, TIA and death), cognitive decline, or a new brain infarction. Candidate predictors include age, gender, side of stenosis, symptomatic stenosis, time from symptoms to CEA, percentage of ipsilateral ICA stenosis, percentage of contralateral ICA stenosis, arterial hypertension, diabetes mellitus, hyperlipidemia, smoking, alcohol abuse, coronary heart disease, atrial fibrillation, type of anesthesia, shunt use, antithrombotic drug use, number of antihypertensive drugs, insulin use, oral antidiabetics use, perioperative use of heparin, perioperative dose of heparin, statin use, dose of statin, type of plaque in ipsilateral carotid stenosis. All models will include the treatment group. Results will be reported as odds ratio with 95% CI.

Data will be analyzed using R (R Development Core Team. 2008. R: A language and environment for statistical computing. R Foundation for Statistical Computing. Vienna, Austria), Stata (StataCorp. 2017. Stata Statistical Software: Release 15. College Station, TX: StataCorp LLC) and/or SPSS (IBM, Armonk, NY, USA).

ELIGIBILITY:
Inclusion Criteria:

* Subject has a symptomatic or asymptomatic ICA stenosis ≥ 70 % (NASCET criteria) as detected by a duplex sonography (see Appendix) and confirmed using the computed tomography angiography (CTA), magnetic resonance angiography (MRA) or digital subtraction angiography (DSA).
* Subject is indicated for CEA according to the criteria set by the American Heart Association.
* Subject is aged 40 - 85 years.
* Subject has a sufficient temporal bone window for TCD with detectable blood flow in the MCA.
* Subject is functionally independent with a modified Rankin score value of 0 - 2 points.
* Informed consent is signed by the subject.

Exclusion Criteria:

* Subject has been participating in another clinical trial within last 6 weeks.
* Subject has any other medical condition that would make him/her inappropriate for study participation, in the Investigator opinion.

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1492 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2022-11 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
Occurence of ischemic stroke, transient ischemic attack and death within 30 days | 30 days after randomization
  The incidence of ischemic stroke, transient ischemic attack and death within 30 days in sonolysis and control groups

SECONDARY OUTCOMES:
Occurrence of death within 30 days | 30 days after randomization
  The incidence of death within 30 days, collected from the family members and/or from electronic hospital database and/or health insurance companies databases
Occurrence of death within 1 year | 30 year after randomization
  The incidence of death within 1 year, collected from the family members and/or from electronic hospital database and/or health insurance companies databases
Occurrence of any stroke within 30 days | 30 days after randomization
  The incidence of any stroke within 30 days, including 1/ cerebral ischemic stroke defined as acute focal neurological dysfunction caused by focal infarction at single or multiple sites of the brain or retina with evidence coming either from symptoms duration lasting more than 24 h and neuroimaging or other technique in the clinically relevant area or the brain; 2/ intracerebral hemorrhage defined as acute neurological dysfunction caused by hemorrhage within the brain parenchyma or in the ventricular system; 3/ subarachnoid hemorrhage defined as acute neurological dysfunction caused by subarachnoid hemorrhage; 4/ stroke not known if ischemic or hemorrhagic defined as acute focal neurological dysfunction lasting more than 24 hours (or lead to death in less than 24 hours), but subtype of stroke (ischemic or hemorrhagic) has not been determined by neuroimaging or other techniques.
Occurrence of myocardial infarction within 30 days | 30 days after randomization
  The incidence of myocardial infarction within 30 days, defined as post-interventional cardiac troponin T level increase > 2 times the normal upper limit in addition to either chest pain, symptoms consistent with heart ischemia, or electrocardiographic evidence of ischemia
Changes in cognitive functions within 1 year | 1 year after randomization
  Changes in cognitive functions measured by Addenbrooke's Cognitive Examination Revised (ACE-R) at 1 year (at visit 5) compared to baseline (at visit 2)
Changes in cognitive functions within 30 days | 30 days after randomization
  Changes in cognitive function measured by Addenbrooke's Cognitive Examination Revised (ACE-R) 30 days after randomization (at visit 4) compared to baseline (at visit 2)
Postprocedural changes in cognitive functions | 24 hours after intervention
  Changes in cognitive function measured by Addenbrooke's Cognitive Examination Revised (ACE-R) 24 hours after CEA (at visit 3) compared to baseline (at visit 2)
Occurence of new ischemic lesion on post-procedural brain DWI-MRI (Substudy) | 24 hours after intervention
  Appearance of at least one new ischemic lesion on post-procedural brain MR (24 hours after CEA, visit 3), defined as hyperintense region on post-intervention DWI that was not present on pre-treatment images (visit 1).
Number of new ischemic lesions on brain DWI-MRI (Substudy) | 24 hours after intervention
  Number of new ischemic lesions on post-procedural brain MR (24 hours after CEA, visit 3), defined as hyperintense regions on post-intervention DWI that were not present on pre-treatment images (visit 1).
Occurence of new ischemic lesion ≥0.5 mL on post-procedural brain DWI-MRI (Substudy) | 24 hours after intervention
  Appearance of at least one new ischemic lesion ≥0.5 mL on post-procedural brain DWI-MR (24 hours after CEA, visit 3), defined as hyperintense regions on post-intervention DWI that were not present on pre-treatment images (visit 1) with total infarct volume ≥0.5 mL. The volume of new brain infarctions will be measured manually. Infarct volumes will be calculated as the total hyperintense area in single slices multiplied by an effective slice thickness [(actual slice thickness + distance factor)/interslice gap].
Occurence of new ipsilateral ischemic lesion on post-procedural brain DWI-MRI (Substudy) | 24 hours after intervention
  Appearance of at least one new ipsilateral ischemic lesions on post-procedural brain DWI-MR (24 hours after CEA, visit 3), defined as hyperintense regions on post-intervention DWI in the territory of intervened internal carotid artery that were not present on pre-treatment images (visit 1).
Occurence of hemorrhagic stroke | 30 days after randomization
  Incidence of hemorrhagic stroke including subarachnoid hemorrhage within 30 days
Occurence of intracranial bleeding (including brain microbleeds) on control T2*-MR (substudy) | 24 hours after intervention
  Incidence of intracranial bleeding (including brain microbleeds) on control T2*-MR in the MR substudy

OTHER OUTCOMES:
Occurence of new ischemic lesions on brain DWI-MRI (Substudy) | 24 hours after intervention
  The incidence of new ischemic lesions on brain DWI-MRI performed 24 hours after the CEA in sonolysis and control groups - Primary outcome for the Substudy
Occurence of new ischemic lesions on brain DWI-MRI in local anesthesia and general anesthesia (Substudy) | 24 hours after intervention
  The incidence of new ischemic lesions on brain DWI-MRI performed 24 hours after the CEA in patients with surgery in local anesthesia and general anesthesia
Cosmetic outcome in patients after carotid endarterectomy using short longitudinal and transverse skin incision (Substudy) | 3 months after intervention
  The total score in the Patient and Observer Scar Assessment Scale in patients after carotid endarterectomy using short longitudinal and transverse skin incision (Substudy)
Changes in Mini Mental State Examination (MMSE) within 1 year | 1 year after randomization
  Changes in cognitive functions measured by MMSE at 1 year (at visit 5) compared to baseline (at visit 2)
Changes in Mini Mental State Examination (MMSE) within 30 days | 30 days after randomization
  Changes in cognitive functions measured by MMSE at 30 days after randomization (at visit 4) compared to baseline (at visit 2)
Postprocedural changes in Mini Mental State Examination (MMSE) | 24 hours after CEA
  Changes in cognitive functions measured by MMSE at 24 hours after CEA (at visit 3) compared to baseline (at visit 2)
Changes in Clock Drawing Test within 1 year | 1 year after randomization
  Changes in cognitive functions measured by Clock Drawing Test at 1 year (at visit 5) compared to baseline (at visit 2)
Changes in Clock Drawing Test within 30 days | 30 days after randomization
  Changes in cognitive functions measured by Clock Drawing Test at 30 days after randomization (at visit 4) compared to baseline (at visit 2)
Postprocedural changes in Clock Drawing Test | 24 hours after CEA
  Changes in cognitive functions measured by Clock Drawing Test at 24 hours after CEA (at visit 3) compared to baseline (at visit 2)
Changes in Speech Fluency Test within 1 year | 1 year after randomization
  Changes in cognitive functions measured by Speech Fluency Test at 1 year (at visit 5) compared to baseline (at visit 2)
Changes in Speech Fluency Test within 30 days | 30 days after randomization
  Changes in cognitive functions measured by Speech Fluency Test at 30 days after randomization (at visit 4) compared to baseline (at visit 2)
Postprocedural changes in Speech Fluency Test | 24 hours after CEA
  Changes in cognitive functions measured by Speech Fluency Test at 24 hours after CEA (at visit 3) compared to baseline (at visit 2)

CONTACTS AND LOCATIONS:
Overall Officials: David Skoloudik, MD,PhD,FESO, Study Chair — Department of Neurology, University Hospital Ostrava
Locations (1):
- University Hospital Ostrava, Ostrava, Czech Republic, Czechia

IPD SHARING:
Plan to Share IPD: Yes
The IPD sharing plan will be created prior to publication of study results.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The data will become available after publication for 10 years.
Access Criteria: The IPD sharing access criteria will be created prior to publication of study results.

REFERENCES:
- [Background] Hrbac T, Netuka D, Benes V, Nosal V, Kesnerova P, Tomek A, Fadrna T, Benes V Jr, Fiedler J, Priban V, Brozman M, Langova K, Herzig R, Skoloudik D. SONOlysis in prevention of Brain InfaRctions During Internal carotid Endarterectomy (SONOBIRDIE) trial - study protocol for a randomized controlled trial. Trials. 2017 Jan 17;18(1):25. doi: 10.1186/s13063-016-1754-x. PMID 28095924
- [Derived] Skoloudik D, Hrbac T, Kovar M, Benes V 3rd, Fiedler J, Branca M, Rossel JB, Netuka D; SONOBIRDIE Trial Investigators. Sonolysis during carotid endarterectomy: randomised controlled trial. BMJ. 2025 Mar 19;388:e082750. doi: 10.1136/bmj-2024-082750. PMID 40107675
- [Derived] Orlicky M, Hrbac T, Sames M, Vachata P, Hejcl A, Otahal D, Havelka J, Netuka D, Herzig R, Langova K, Skoloudik D. Anesthesia type determines risk of cerebral infarction after carotid endarterectomy. J Vasc Surg. 2019 Jul;70(1):138-147. doi: 10.1016/j.jvs.2018.10.066. Epub 2019 Feb 18. PMID 30792052